CLINICAL TRIAL: NCT01257438
Title: Prospective, Multi-Center, Randomized, Concurrently-Controlled Study of the FLUENCY® PLUS Endovascular Stent Graft in the Treatment of In-stent Restenosis in the Arteriovenous (AV) Access Venous Outflow Circuit (RESCUE)
Brief Title: FLUENCY® PLUS Endovascular Stent Graft for In-stent Restenosis
Acronym: RESCUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPV-08-002
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluency Plus Endovascular Stent Graft (Experimental): Fluency Plus Endovascular Stent Graft
  Interventions: Device: Fluency Plus Endovascular Stent Graft
- Percutaneous Transluminal Angioplasty (Active Comparator): Percutaneous Transluminal Angioplasty only
  Interventions: Device: Percutaneous Transluminal Angioplasty only

INTERVENTIONS:
Device: Fluency Plus Endovascular Stent Graft — Treatment of in-stent restenosis
  Arms: Fluency Plus Endovascular Stent Graft
Device: Percutaneous Transluminal Angioplasty only — Treatment of in-stent restenosis
  Arms: Percutaneous Transluminal Angioplasty

SUMMARY:
The primary purpose of this study is to demonstrate that the FLUENCY® PLUS Endovascular Stent Graft can effectively and safely treat in-stent restenotic lesions in the venous outflow of the Arteriovenous (AV) access circuit of hemodialysis patients with either of the two predominant vascular access types - those with an AV graft and those with an AV fistula.

DETAILED DESCRIPTION:
This study will compare the use of the FLUENCY® PLUS Endovascular Stent Graft (following Percutaneous Transluminal Angioplasty (PTA)) to PTA alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient must voluntarily sign and date the Informed Consent Form (ICF) prior to collection of study data or performance of study procedures.
* Patient must be either a male or non-pregnant female ≥ 21 years of age with an expected lifespan sufficient to allow for completion of all study procedures.
* Patient must be willing to comply with the protocol requirements, including the follow-up procedures, and be contacted by telephone.
* Patient must have an AV access graft (implanted for ≥ 30 days) or mature fistula located in an arm, and must have undergone at least one successful dialysis session prior to the index procedure.
* Patient must have a previously-placed bare metal stent located in the venous outflow of the AV access circuit in which a ≥ 50% stenosis originates.
* The entire target lesion must be located in the restenosed bare metal stent and extend to no more than 3 cm outside of the bare metal stent.
* The target lesion must be ≤ 10 cm in length.
* After angiography, the operator must judge that the lesion is amenable to angioplasty.
* The reference vessel diameter at the restenosed bare metal stent must be between 5.0 mm and 12.0 mm.
* Additional stenotic lesions (≥ 50%) in the venous outflow that are > 3cm from the edge of the target lesion must be successfully treated (defined as < 30% residual stenosis) prior to the index procedure.

Exclusion Criteria:

* The target lesion has had a corresponding thrombosis treated within 7 days prior to the index procedure.
* The target lesion has a reference vessel diameter that is larger than 12.0 mm.
* The patient has an infected AV access graft/fistula or uncontrolled systemic infection.
* A pseudoaneurysm is present within the target lesion.
* The location of the target lesion would require that the FLUENCY® PLUS Endovascular Stent Graft be deployed across the elbow joint.
* The location of the target lesion would require that the FLUENCY® PLUS Endovascular Stent Graft be deployed at or across the segment of graft or fistula utilized for dialysis needle puncture (i.e., "cannulation zone").
* The location of the target lesion would require that the FLUENCY® PLUS Endovascular Stent Graft cross the cephalic arch (perpendicular portion of the cephalic vein in the region of the deltopectoral groove before its junction with the axillary vein).
* The location of the target lesion would require that the FLUENCY® PLUS Endovascular Stent Graft be placed in the Superior Vena Cava.
* The location of the target lesion would require that the FLUENCY® PLUS Endovascular Stent Graft is placed across an angle that is greater than 90 degrees.
* The restenosed bare metal stent is fractured, as verified by angiography per institution's standard of care.
* The patient has a known uncontrolled blood coagulation disorder.
* The patient has a known allergy or sensitivity to contrast media which cannot be adequately pre-medicated.
* The patient has a known hypersensitivity to nickel-titanium.
* The subject has another medical condition, which, in the opinion of the Investigator, may cause him/her to be non-compliant with the protocol, confound the data interpretation, or is associated with a life expectancy insufficient to allow for the completion of study procedures and follow-up.
* The patient is currently participating in an investigational drug or another device study that has not completed the study treatment or that clinically interferes with the study endpoints. Note: Studies requiring extended follow-up visits for products that were investigational, but have since become commercially available, are not considered investigational studies.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2010-12; Primary Completion 2013-11 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Falk, M.D., Principal Investigator — Access Center of New Jersey; Ivan Maya, MD, Principal Investigator — Nephrology Associates of Central Florida; Alexander Yevzlin, MD, Principal Investigator — University of Wisconsin, Madison
Locations (23):
- United States (23):
  - University of Alabama Radiology Dept, Birmingham, Alabama
  - Southwest Kidney Institute Inc, Phoenix, Arizona
  - Arizona Kidney Disease & Hypertension Center-Surgery Center, Phoenix, Arizona
  - Capital Nephrology Access Center, Sacramento, Arizona
  - Angiocare LLC w/Renal Care Associates PC, Tucson, Arizona
  - Greater Long Beach Vascular Access Center, Bellflower, California
  - Ladenheim Dialysis Access Centers, Fresno, California
  - American Access Care Connecticut Image Guided Surgery, Fairfield, Connecticut
  - Yale University, New Haven, Connecticut
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Vascular & Interventional Care Center, Augusta, Georgia
  - Savannah Vascular Surgery, Savannah, Georgia
  - MakrisMD, LLC, d/b/a Chicago Access Care, Hinsdale, Illinois
  - The Vascular Access Center, West Springfield, Massachusetts
  - ProHEALTH Care Associates LLP, Lake Success, New York
  - Capital Access Center, Raleigh, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Access Care, Providence, Rhode Island
  - Premeire Vascular Access and Imaging Center, Knoxsville, Tennessee
  - Renal Associates, P.A. Research Division, San Antonio, Texas
  - American Access Care of Richmond, Richmond, Virginia
  - University of Wisconsin School of Medicine & Public Health, Madison, Wisconsin
  - Midwest Nephrology Associates Vascular Access Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluency: Fluency Plus Endovascular Stent Graft
  Fluency Plus Endovascular Stent Graft: Treatment of in-stent restenosis
- PTA Only: PTA only: Treatment of in-stent restenosis
Period: Overall Study
Arm/Group | Fluency | PTA Only
Started | 132 | 143
Completed | 102 | 97
Not Completed | 30 | 46

BASELINE CHARACTERISTICS:
Population: 275 subjects were enrolled but, the primary effectiveness endpoint was statistically tested with 220 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluency | PTA Only | Total
Number analyzed (Participants) | 132 | 143 | 275
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (13.57) | 61.1 (13.47) | 61.9 (13.52)
Gender [Count of Participants; unit: Participants]
  Female | 64 | 70 | 134
  Male | 68 | 73 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 18 | 39
  Not Hispanic or Latino | 111 | 125 | 236
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 4 | 4
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 72 | 84 | 156
  White | 57 | 50 | 107
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 132 | 143 | 275

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Access Circuit Primary Patency (ACPP) That is Superior for FLUENCY® PLUS Endovascular Stent Graft (Following Percutaneous Transluminal Angioplasty (PTA)) Over PTA Alone Through Six Months.
Description: Access Circuit Primary Patency (ACPP) is defined as the interval following the index intervention until the next access thrombosis or repeated intervention. ACPP ends with a reintervention anywhere within the access circuit, from the arterial inflow to the superior vena cava-right atrial junction. Venous rupture caused by PTA is not an ACPP failure unless achieving hemostasis also causes thrombosis. Freedom from access thrombosis or repeated intervention is the criteria for success.
Time Frame: 6 months
Population: Subjects at risk (at 6 months) is a calculation in Kaplan-Meier time-to-event analyses that refers to subjects who have not had ACPP failure through the 6 months (i.e., are event-free through 6 months).
Measure: Number (95% Confidence Interval); unit: % of subjects with successful ACPP
Arm/Group | Fluency | PTA Only
Number analyzed (Participants) | 109 | 111
% of subjects with successful ACPP | 16.7 [9.24 to 24.16] | 3.0 [0.00 to 6.27]
Statistical Analysis 1: Comparison: Fluency vs PTA Only; Subjects at risk (at 6 months) is a calculation in Kaplan-Meier time-to-event analyses that refers to subjects who have not had ACPP failure through the 6 months (i.e., are event-free through 6 months); Test type: Superiority or Other; p < 0.001, Log Rank; Greenwood's estimate of variance = 0.59, 95% CI 2-sided [0.44 to 0.79]

2. Primary Outcome: Non-inferiority of FLUENCY® PLUS Endovascular Stent Graft (Following PTA) Over PTA Alone Through 30 Days in the Treatment of In-stent Restenotic Lesions.
Description: Safety rates measured for the randomized subjects population (both Arteriovenous (AV) Graft and Fistula subjects combined), the percentage of subjects free from safety events through 30 days.
Time Frame: 30 days
Population: Safety rates measured for the randomized subjects population (both AV Graft and Fistula subjects combined), the percentage of subjects free from safety events through 30 days.
Measure: Number (95% Confidence Interval); unit: % of subjects free from safety events
Arm/Group | Fluency | PTA Only
Number analyzed (Participants) | 132 | 143
% of subjects free from safety events | 96.9 [92.31 to 99.16] | 96.4 [91.81 to 98.82]
Statistical Analysis 1: Comparison: Fluency vs PTA Only; Test type: Non-Inferiority or Equivalence — The p-value is based on a non-inferiority Farrington and Manning Exact Test. The non-inferiority margin is 0.075 (or 7.5%); p = 0.007, Farrington and Manning Exact Test; The non-inferiority margin is 0.075 (or 7.5%)

3. Secondary Outcome: Percentage of Participants With Primary Lesion Patency (PLP) That is Superior for FLUENCY® PLUS Endovascular Stent Graft (Following PTA) Over PTA Alone Through Six Months in the Treatment of In-stent Restenotic Lesions.
Description: Primary Lesion Patency (PLP) is defined as the interval after the index intervention until the next re-intervention at the original treatment site or until the extremity is abandoned for permanent access. Freedom from re-intervention is the criteria for success.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: % of subjects with successful PLP
Arm/Group | Fluency | PTA Only
Number analyzed (Participants) | 109 | 111
% of subjects with successful PLP | 65.2 [55.59 to 74.86] | 10.4 [4.30 to 16.57]

ADVERSE EVENTS:
Time Frame: all adverse events involving the AV access circuit that were reported by the Investigators from index procedure onward through 6 months, regardless of whether or not the events were classified by the Clinical Events Committee (CEC) as safety events.
Arm/Group | Fluency | PTA Only
Serious Adverse Events (participants affected / at risk) | 4/128 | 4/137
Other Adverse Events (participants affected / at risk) | 11/128 | 8/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluency (N=128) | PTA Only (N=137)
Infection in the AVF venous cannulation site (Infections and infestations) | 1 (1) | 1 (1)
infection of the old stent in the fistula (Infections and infestations) | 1 (1) | 0 (0)
vessel rupture (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
arm or hand edema (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
rash on arm due to allergic reaction to unknown source (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
fever/cellulitis of both legs/sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluency (N=128) | PTA Only (N=137)
Hemorrhage (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 2 (2)
Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arm or Hand Edema (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pseudoaneurysm (Vascular disorders) | 2 (2) | 0 (0)
Vessel Rupture (Vascular disorders) | 0 (0) | 2 (2)
Allergic reaction. to uncertain source; rash on right arm (Infections and infestations) | 1 (1) | 0 (0)
Fever/cellulitis of both legs/sepsis (Infections and infestations) | 1 (1) | 0 (0)
Infolded covered stent (Vascular disorders) | 0 (0) | 1 (1)
Prolonged Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
hemoptysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other